CLINICAL TRIAL: NCT01810354
Title: PROPHYLACTIC ANTIBIOTICS PRIOR TO CESAREAN SECTION IN OBESE WOMEN: Does Increasing the Dose Increase the Tissue Concentration?
Brief Title: PROPHYLACTIC ANTIBIOTICS PRIOR TO CESAREAN SECTION IN OBESE WOMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Lindsay Maggio,, Maternal-Fetal Medicine Fellow, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-0004
Record Dates: First submitted 2013-03-07; First posted 2013-03-13 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Infection Prevention
Keywords: Cefazolin; Tissue concentration; infection; cesarean section; obese
MeSH Terms: conditions — Infections; Obesity | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two grams cefazolin (Experimental): Two grams of cefazolin will be given by intravenous bolus zero to 60 minutes prior to the start of the cesarean section.
  Interventions: Drug: Cefazolin
- Three grams cefazolin (Active Comparator): Three grams of cefazolin will be given by intravenous bolus zero to 60 minutes prior to the start of the cesarean section.
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin

SUMMARY:
Surgical site infections are common and a cause of major morbidity. They are also more common in obese women. Cesarean sections are the most common surgery performed in the United States, therefore pregnant women are being faced with this problem frequently. There is evidence to show that prophylactically administered antibiotics, cefazolin specifically, to obese women prior to cesarean section do not reach adequate concentrations in adipose tissue to prevent infection. The purpose of this study is to evaluate if an increased dose of cefazolin will attain adequate tissue concentration in obese women. Our hypothesis is that three grams of cefazolin given no more than 60 minutes prior to the start of a cesarean section in an obese (Body mass index (BMI) greater than or equal to 30) woman will attain adequate adipose tissue concentration compared to two grams of cefazolin.

Subjects will be selected if they are greater than 37 weeks gestation wiht a singleton pregnancy and require a cesarean section for any obstetrical indication. Women will be excluded if they have a suspected infection, have a multiple gestation, or have preexisting diabetes or hypertension with end organ damage. The subjects will be screened both by through the OR schedule as well as through the clinics. They will then be consented and enrolled by the primary investigator. Once enrolled the subjects will be randomized to receive either two grams or three grams of cefazolin as prophylactic antibiotics to be given no more than 60 minutes prior to the start of the surgery.

Two adipose tissue samples will be obtained at the time of surgery. The first at the start after skin incision and the second at the end prior to closure of the skin. There will also be a separate IV placed at the start of the procedure from which three blood draws can be collected. These three samples will be obtained at the start of the surgery but after antibiotic administration, at the time of the first adipose collection, and at the time of the second adipose collection. The samples will then be stored at -80 degrees and shipped to David P. Nicolau's lab in Hartford, CT for the tissue and serum analysis.

While the subjects are in the hospital recovering from their surgery, a chart review will be performed to determine if there are any infections occuring post-operatively. A telephone survey will be conducted six to eight weeks postpartum again assessing for any infectious complications after the cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Obese - body mass index (BMI) calculated as weight (kg)/ [height (m2)]greater than or equal to 30 as determined at their first prenatal visit
* Gestational age of 37 0/7 weeks and greater
* Singleton Pregnancy
* Non-emergent cesarean section

Exclusion Criteria:

* Known cephalosporin allergy
* Severe allergy to penicillin making cephalosporin use a contraindication
* Exposure to antibiotics in the preceding 7 days
* Need for emergent cesarean section
* Multiple gestations
* Suspected chorioamnionitis
* Pre-gestational diabetes
* Chronic hypertension with evidence of end organ damage

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Adipose tissue concentration of cefazolin | At the start of the cesarean section and at the end of the cesarean section
  Two separate two gram samples of adipose tissue will be removed from the subcutaneous tissue. The first sample will be removed after skin incision, yet prior to fascial incision. The second sample will be collected after fascial closure, yet prior to skin closure.

SECONDARY OUTCOMES:
Serum cefazolin concentrations | After antibiotic infusion, at the start of the cesarean section, and at the end of the cesarean section
  Three separate intraoperative blood samples will be collected to evaluate the serum cefazolin concentrations. The first sample will be collected after antibiotic administration, prior to the surgery start. The next two samples will be collected coincidental to the time of adipose tissue collection. The first after skin incision, yet prior to fascial incision. The second after fascial closure, yet prior to skin closure.

OTHER OUTCOMES:
Infectious morbidity | Participants will be followed for a duration of 6-8 weeks after the cesarean section
  While in the hospital, chart reviews of the subject will be performed to identify any infectious complications. A follow-up telephone survey will be conducted to assess for this outcome as well at six to eight weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Maggio, MD, Principal Investigator — Women & Infant's Hospital; Brenna Anderson, MD, Study Director — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Maggio L, Nicolau DP, DaCosta M, Rouse DJ, Hughes BL. Cefazolin prophylaxis in obese women undergoing cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2015 May;125(5):1205-1210. doi: 10.1097/AOG.0000000000000789. PMID 25932849